CLINICAL TRIAL: NCT01845142
Title: Immunologic Functions of a Single Dose of 100.000 I.U. Cholecalciferol (Vitamin D3)
Brief Title: Immunologic Action of a Single Dose Cholecalciferol
Acronym: ViDImmun
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Margitta Worm (Other)
Responsible Party: Sponsor-Investigator, Margitta Worm, Prof. Dr. med., Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: ViDImmun; 2012-003217-33 (EudraCT Number)
Record Dates: First submitted 2013-04-24; First posted 2013-05-03 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D; vitamin D deficiency; immune cells; pharmacokinetic; < 50 nmol/L 25(OH)D serum concentration
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- intramuscular 100.000 I.U. vitamin D3 (Active Comparator): intramuscular 100.000 I.U. vitamin D3
  Interventions: Drug: single administration of 100.000 I.U. vitamin D
- intramuscular placebo (Placebo Comparator): intramuscular 0.9% sodium chloride
  Interventions: Drug: Placebo
- subcutaneous 100.000 I.U. vitamin D3 (Active Comparator): subcutaneous 100.000 I.U. vitamin D3
  Interventions: Drug: single administration of 100.000 I.U. vitamin D
- subcutaneous placebo (Placebo Comparator): subcutaneous 0.9% sodium chloride
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: single administration of 100.000 I.U. vitamin D
  Other Names: cholecalciferol
  Arms: intramuscular 100.000 I.U. vitamin D3; subcutaneous 100.000 I.U. vitamin D3
Drug: Placebo
  Arms: intramuscular placebo; subcutaneous placebo

SUMMARY:
Vitamin D receptors are expressed in activated different immune cells. It is not known, which immune cell type is targeted by exogenous vitamin D. Here, vitamin D-deficient individuals will receive once 100.000 I.U. vitamin D3 either intramuscular or subcutaneous in a double-blind placebo controlled setting. Immune cells will be monitored from the blood over time.

DETAILED DESCRIPTION:
Vitamin D-deficient individuals will receive once

* double-blind, placebo controlled 100.000 I.U.vitamin D3
* intramuscular or subcutaneous

Blood will be taken over time and

* immune cells (T cells, B cells, myeloid antigen presenting cells) are characterized by flow-cytometry
* vitamin D-metabolites will be monitored

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* 18-60 yrs
* 25-hydroxyvitamin D serum below 50 nmol/L
* women only: effective contraception

Exclusion Criteria:

* 25-hydroxyvitamin D serum above 50 nmol/L
* body-mass index <18 or >30 kg per m2
* planned UV-exposure (UV-index > 5)
* hypersensitivity to vitamin D
* history of hypercalcemia, kidney stones, kidney insufficiency, sarcoidosis, pseudohyperparathyroidism concomitant vitamin A- and/or vitamin D treatment
* treatment with immunosuppressants, immunomodulators, phenytoin, barbiturate, thiazide-diuretics, glycosides
* immobile patients
* out of normal range on screening visit (calcium,phosphate,creatinin,hematology)
* psychiatric hospitalization
* pregnancy / breast-feeding
* dependency / relationship on sponsor
* concomitant participation in other clinical trials (30 days before)
* drug or alcohol abuse
* lack of compliance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in the numbers of vitamin D-responsive B cells after vitamin D administration. | up to 3 months
  Peripheral B cells will be isolated before, after 1 week, 1 month and 3 months after vitamin D administration and characterized by flow-cytometry. Vitamin D-responsive B cells will be quantified before and 1 week, 1 month and 3 months after vitamin D administration.

SECONDARY OUTCOMES:
Characterize vitamin D-responding myeloid immune cells | up to 3 months
  peripheral blood mononuclear cells will be isolated before, after 1 week, 1 month and 3 months after vitamin D administration and monocytes will be characterized phenotypically by flow-cytometry.
Impact of vitamin D on specific humoral memory | up to 3 months
  The humoral immunoglobulin response against selected endogenous viruses (anti-virus-specific-Ig) over time will be determined before and 3 months after vitamin D administration.
Vitamin D pharmacokinetics | up to 3 months
  Vitamin D-metabolites including 25-hydroxyvitamin D will be determined up to 3 months after administration of a single dose-vitamin D.
Characterize vitamin D-responsive T cells | up to 3 months
  peripheral T cells will be isolated before, after 1 week, 1 month and 3 months after vitamin D administration and characterized by flow-cytometry according to functional subpopulations.

CONTACTS AND LOCATIONS:
Overall Officials: Margitta Worm, Prof, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Dpt of Dermatology and Allergology, Charité University Medicine Berlin, Berlin, State of Berlin, Germany